CLINICAL TRIAL: NCT06415578
Title: Effectiveness of Ergonomics Training and Exercise in Esports Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar9
Record Dates: First submitted 2024-05-09; First posted 2024-05-16 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Musculoskeletal Diseases; Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Diseases; Musculoskeletal Pain | interventions — Ergonomics; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): Only ergonomics training will be given
  Interventions: Other: ergonomics training
- exercise (Experimental): Exercise training will be provided along with ergonomics training.
  Interventions: Other: ergonomics training; Other: Exercises

INTERVENTIONS:
Other: ergonomics training — In this training; What is ergonomics, the importance of ergonomics, the purpose of ergonomics, risk factors for musculoskeletal disorders that can be seen in e-sports players, ergonomic arrangements that can be made in the working environment and methods of protection from musculoskeletal injuries, posture disorders and various ergonomic arrangements that can be made for posture disorders and chair selection, screen selection. selection and rest breaks were included. Participants will be trained twice in total, on the first day of the study and at the end of the 4th week. The training will be carried out interactively, supported by videos and visuals. Training will be done individually and will last approximately 2 hours.
Other: Exercises — The exercise training program will be implemented for 8 weeks, 3 days a week, lasting an average of 45 minutes. All participants will be given information about the exercises before the exercise training. The exercise protocol was designed as 3 parts: warm-up, exercise and cool-down. Stretching exercises, mobility and strength exercises will be applied. A rest period of 30-45 seconds was given between sets and 2-3 minutes between exercises. Participants will be given dynamic and static stretching, nerve stretching, postural strength and functional exercises for the upper extremity. Relevant movements will be modified according to the exercise capacity of the participants. Exercise content will also include median, ulnar and radial nerve stretching, neck and thoracic mobility exercises, and functional strength exercises for the shoulder, arm, hand and wrist. Exercise tracking will be checked regularly through online conversations.
  Arms: exercise

SUMMARY:
The aim of this study is to investigate the effectiveness of ergonomics training and exercise in e-sports players.

DETAILED DESCRIPTION:
After detailed information about the study is given to the individuals to be included in the study, individuals who voluntarily agree to participate in the study will sign an informed consent form. Participants will be divided into 2 groups consisting of equal numbers of individuals. The groups were called control group and exercise group. All participants will be given ergonomics training. In addition to the exercise group, exercise training will be given for 8 weeks, 3 days a week and 45 minutes a day. Sociodemographic information form, Arm, Shoulder and Hand Problems Questionnaire (DASH), Neck Disability Questionnaire (NDI), Rapid Upper Extremity Assessment (RULA) and Pittsburgh Sleep Quality Index (PSQI) will be used as evaluation scales. Evaluations will be made at the beginning and end of the study. will be done once.

ELIGIBILITY:
Inclusion Criteria:

* those who signed the voluntary consent form
* Having actively participated in E-sports organizations and tournaments within 16 months
* not having a chronic disease that will affect the musculoskeletal system
* Not having any health problems that prevent him from exercising and not having had a surgical operation in the last 6 months.

Exclusion Criteria:

* Players under 18 years of age
* have a chronic disease that affects the musculoskeletal system
* Having had a surgical operation in the last 6 months that would prevent him from being interested in e-sports games

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 8 weeks
  This index evaluates sleep quality and disturbance over the past month. It contains a total of 24 questions. 19 of these questions are answered by the person's self-assessment, and 5 of them are answered by the roommate who shares the same room with the person. The 5 questions answered by the person's roommate are not included when calculating the score. In scoring, the lowest (0) and the highest (21) points are obtained. A score of 4 and above indicates poor sleep quality.
Rapid Upper Limb Assessment | 8 weeks
  It is an ergonomics risk assessment method that quickly analyzes the employee's upper extremity from an ergonomic perspective. It evaluates upper extremity movements in 14 separate steps. 8 of these steps are scored for arm and hand position, and 6 for neck and trunk position, according to the table. The minimum Rapid Upper Limb Assessment Score = 1, and the maximum Rapid Upper Limb Assessment Score = 7. A high score means high risk.
Disabilities of the Arm, Shoulder and Hand Questionnaire | 8 weeks
  It was developed to evaluate functional status and symptoms by focusing on physical function in upper extremity injuries. According to the results of the survey; a result from 0-100 is obtained from each part; 0-no apology 100-maximum apology.
Neck disability index | 8 weeks
  There are 10 parameters in the Neck disability index, each with 6 answer choices. These; The severity of neck pain is personal care, lifting loads, reading, headache, concentration, business life, driving, sleep and leisure activities. It is scored between 0 (no pain or functional limitation) and 5 (maximum pain and maximum limitation). The subjects were asked to choose the most appropriate option for themselves from each parameter. At the end of the survey, the total score was determined by adding up the scores of the selected options. In the Neck disability index, 35 points and above were defined as complete apology, 25 to 34 points as severe apology, 15 to 24 points as moderate apology, 5 to 14 points as mild apology, and 0 to 4 points as no apology.

CONTACTS AND LOCATIONS:
Overall Officials: Atakan GÜRGAN, Study Chair — Uskudar University
Locations (1):
- Uskudar Üniversity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monteiro Pereira A, Costa JA, Verhagen E, Figueiredo P, Brito J. Associations Between Esports Participation and Health: A Scoping Review. Sports Med. 2022 Sep;52(9):2039-2060. doi: 10.1007/s40279-022-01684-1. Epub 2022 Apr 29. PMID 35486374
- [Background] Ketelhut S, Martin-Niedecken AL, Zimmermann P, Nigg CR. Physical Activity and Health Promotion in Esports and Gaming-Discussing Unique Opportunities for an Unprecedented Cultural Phenomenon. Front Sports Act Living. 2021 Sep 16;3:693700. doi: 10.3389/fspor.2021.693700. eCollection 2021. PMID 34604743
- [Background] DiFrancisco-Donoghue J, Balentine J, Schmidt G, Zwibel H. Managing the health of the eSport athlete: an integrated health management model. BMJ Open Sport Exerc Med. 2019 Jan 10;5(1):e000467. doi: 10.1136/bmjsem-2018-000467. eCollection 2019. PMID 30792883
- [Background] Seffah KD, Salib K, Dardari L, Taha M, Dahat P, Toriola S, Satnarine T, Zohara Z, Adelekun A, Ahmed A, Gutlapalli SD, Patel D, Khan S. Health Benefits of Esports: A Systematic Review Comparing the Cardiovascular and Mental Health Impacts of Esports. Cureus. 2023 Jun 20;15(6):e40705. doi: 10.7759/cureus.40705. eCollection 2023 Jun. PMID 37485153
- [Background] Eltayeb SM, Staal JB, Hassan AA, Awad SS, de Bie RA. Complaints of the arm, neck and shoulder among computer office workers in Sudan: a prevalence study with validation of an Arabic risk factors questionnaire. Environ Health. 2008 Jun 27;7:33. doi: 10.1186/1476-069X-7-33. PMID 18588691